CLINICAL TRIAL: NCT00665340
Title: A Randomized, Double Blind, Placebo-controlled, Parallel Group, Multi-center Study to Investigate the Responsiveness of the Erectile Quality Scale (EQS) to Vardenafil HCl Flexible Dose Versus Placebo in Males With Erectile Dysfunction.
Brief Title: Investigate the Responsiveness of the Erectile Quality Scale to Vardenafil Flexible Dose vs Placebo in Males With Erectile Dysfunction (ED)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 11561
Record Dates: First submitted 2008-04-18; First posted 2008-04-23 (Estimated); Last update posted 2013-10-11 (Estimated); Status verified 2013-10

CONDITIONS: Erectile Dysfunction
Keywords: Erectile Dysfunction; Vardenafil
MeSH Terms: conditions — Erectile Dysfunction | interventions — Vardenafil Dihydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Arm 1 (Placebo Comparator)
  Interventions: Drug: Placebo
- Arm 2 (Experimental)
  Interventions: Drug: Levitra (Vardenafil, BAY38-9456)

INTERVENTIONS:
Drug: Placebo — Matching placebo
  Arms: Arm 1
Drug: Levitra (Vardenafil, BAY38-9456) — 5m, 10 mg and 20 mg 1 h prior to sexual intercourse
  Arms: Arm 2

SUMMARY:
This study was conducted to evaluate in adult men with erectile dysfunction (often called impotence), the effect of vardenafil HCl on the quality of their erections. Many men experience occasional erectile problems during their lives. The causes of erectile dysfunction are varied and may be due to physiological or emotional reasons. This study is designed to study the responsiveness of the erection quality scale (EQS) to vardenafil HCl. In this study, vardenafil HCl will be compared to placebo. Placebo is a pill which looks like the real drug but it is not. It contains no active ingredients.

ELIGIBILITY:
Inclusion Criteria:- Males who have had ED for at least six months- Heterosexual relationship.- Males 18 and older. Exclusion Criteria:- Primary hypoactive sexual desire.- History of myocardial infarction, stroke or life-threatening arrhythmia within the prior 6 months.- Stable heterosexual relationship for > 6 month- Other exclusion criteria apply according to the US Product Information

Ages: 18 Years to 64 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 219 (Actual)
Dates: Start 2004-07; Primary Completion 2005-01 (Actual); Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
Erection Quality Scale | Week 8

SECONDARY OUTCOMES:
Erection Quality Scale | Week 4 and 8
International Index of Erectile Function- Erectile Function domain score | Week 4 and 8
Per-subject success rates based on Sexual Encounter Profile, Question 2 | Week 4, 8 Week 8
Safety and tolerability | Week 8
Patient Diary Questions | Weeks 4, 8 Week 8
Global Assessment Question (GAQ) | Weeks 4, 8 of treatment and Week 8
Percentage of subjects achieving back to normal rates of erectile functioning (IIEF-EF > 25) | Week 8-LOCF
Penetration (SEP2) and Maintenance (SEP3) reliability | Week 8-LOCF

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (12):
- United States (12):
  - Phoenix, Arizona
  - Beverly Hills, California
  - Laguna Hills, California
  - Newport Beach, California
  - Aurora, Colorado
  - Trumbull, Connecticut
  - Aventura, Florida
  - Lawrenceville, New Jersey
  - Poughkeepsie, New York
  - Statesville, North Carolina
  - Wilmington, North Carolina
  - Nashville, Tennessee